CLINICAL TRIAL: NCT00228384
Title: GORE VIABAHN Endoprosthesis Versus Bare Nitinol Stent in the Treatment of Long Lesion (>8cm) Superficial Femoral Artery Occlusive Disease
Brief Title: GORE VIABAHN ENDOPROSTHESIS Peripheral Vascular Disease Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SFA 05-03
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Results first posted 2012-05-28 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2012-05

CONDITIONS: Peripheral Vascular Diseases
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gore VIABAHN Endoprosthesis (Active Comparator)
  Interventions: Device: GORE VIABAHN Endoprosthesis
- Bare Nitinol Stent (BNS) (Active Comparator)
  Interventions: Device: Bare Nitinol Stent

INTERVENTIONS:
Device: GORE VIABAHN Endoprosthesis — Implantation
  Other Names: VIABAHN
  Arms: Gore VIABAHN Endoprosthesis
Device: Bare Nitinol Stent — Implantation
  Arms: Bare Nitinol Stent (BNS)

SUMMARY:
To evaluate the performance of the GORE VIABAHN® Endoprosthesis compared to a bare nitinol stent for the treatment of superficial femoral artery (SFA) occlusive disease in long lesions.

DETAILED DESCRIPTION:
This is a multicenter, prospective, randomized study with clinical and radiographic follow-up for three years post-procedure. Approximately one hundred fifty subjects will be enrolled and randomized into one of two study treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Lifestyle-limiting claudication or rest pain.
* Subject (or their legal guardian) has read, understood and provided written informed consent.
* At least 21 years of age.
* Quality of life questionnaires completed.
* Noninvasive lower extremity arterial studies within 45-days prior to study procedure.
* If applicable, staged ipsilateral vascular procedure ≥ 14-days prior to study procedure.
* If applicable, vascular treatment on non-study leg for bilateral claudication ≥ 14-days prior to study procedure.
* Male, infertile female, or female of child bearing potential practicing an acceptable method of birth control with a negative pregnancy test.
* Projected life expectancy of greater than three years.
* The ability to comply with protocol.
* Angiographic and Lesion Requirements meets protocol criteria.

Exclusion Criteria:

* Untreated flow-limiting aortoiliac occlusive disease.
* Any previous stenting or surgery in the target vessel.
* Subjects with arterial lesions requiring treatment with device diameters other than 6, 7, or 8 mm.
* Severe ipsilateral common femoral/profunda disease requiring surgical intervention.
* Femoral or popliteal aneurysm.
* Non-atherosclerotic disease resulting in occlusion.
* Tibial artery disease requiring treatment.
* Prior ipsilateral femoral artery bypass.
* Severe medical comorbidities.
* Popliteal artery vascular access at any time during procedure.
* Antegrade and retrograde vascular access on the same common femoral artery at the time of the SFA intervention.
* Serum creatinine > 2.5 mg/dL within 45 days prior to study procedure.
* Major distal amputation.
* Septicemia.
* Any previously known coagulation disorder.
* Morbid obesity or operative scarring that precludes percutaneous approach (physician's discretion).
* Contraindication to anticoagulation or antiplatelet therapy.
* Known allergies to stent/stent-graft components.
* History of prior life-threatening reaction to contrast agent.
* Currently participating in another clinical research trial.
* Current peritoneal or hemodialysis.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2005-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Ansel, MD, Principal Investigator — Midwest Cardiology; Patrick Geraghty, MD, Principal Investigator — Washington University School of Medicine; Mark Mewissen, MD, Principal Investigator — St. Luke's Medical Center
Locations (15):
- United States (15):
  - Mayo Clinic Phoenix, Phoenix, Arizona
  - Arkansas Heart, Little Rock, Arkansas
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Vascular Surgical Associate, Austell, Georgia
  - Midwest Heart Foundation, Lombard, Illinois
  - Midwest Institute for Minimally Invasive Therapy, Melrose Park, Illinois
  - St Francis Medical Center, Peoria, Illinois
  - St. Johns Hospital/Prairie Education Research, Springfield, Illinois
  - Ochsner Clinic, New Orleans, Louisiana
  - Washington University, St Louis, Missouri
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Midwest Cardiology Research Foundation, Columbus, Ohio
  - Heritage Valley Health Systems, Beaver, Pennsylvania
  - Allegheney General Hospital, Pittsburgh, Pennsylvania
  - St Luke's Medical Center, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Geraghty PJ, Mewissen MW, Jaff MR, Ansel GM; VIBRANT Investigators. Three-year results of the VIBRANT trial of VIABAHN endoprosthesis versus bare nitinol stent implantation for complex superficial femoral artery occlusive disease. J Vasc Surg. 2013 Aug;58(2):386-95.e4. doi: 10.1016/j.jvs.2013.01.050. Epub 2013 May 13. PMID 23676191

RESULTS

PARTICIPANT FLOW:
Groups:
- GORE VIABAHN Endoprosthesis: Subjects randomized to this group received the Gore VIABAHN Endoprosthesis.
- Bare Nitinol Stent: Subjects randomized to this group received a Bare Nitinol Stent (BNS) per the implanting physician's standard of care.
Period: Overall Study
Arm/Group | GORE VIABAHN Endoprosthesis | Bare Nitinol Stent
Started | 72 | 76
Baseline | 72 | 76
30-Day Follow-up (Safety Outcome) | 69 | 72
Three Year Follow-up (Final) | 43 | 47
Completed | 43 | 47
Not Completed | 29 | 29
Not completed — Death | 9 | 3
Not completed — Lost to Follow-up | 6 | 10
Not completed — Surgical Intervention (bypass) | 5 | 5
Not completed — Withdrawal by Subject | 9 | 10
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GORE VIABAHN Endoprosthesis | Bare Nitinol Stent | Total
Number analyzed (Participants) | 72 | 76 | 148
Age Continuous [Median (Full Range); unit: years] | 69 [45 to 90] | 63 [43 to 89] | 67 [43 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 27 | 54
  Male | 45 | 49 | 94
Region of Enrollment [Number; unit: participants]
  United States | 72 | 76 | 148

OUTCOME MEASURES:

1. Primary Outcome: Efficacy: Primary Patency at Three Years
Description: Primary patency is the Peak Systolic Velocity Ratio (PSVR) maintained at or below 2.0 without any repeat intervention.
  The PSVR is the ratio of the highest velocity (or pressure) of the blood moving through the stent divided by the velocity immediately outside the stent (the end of the stent nearest to the heart). Pressures are measured by ultrasound. These results include the percentage of subjects that maintained primary patency at or below 2.0 without any repeat intervention through the end of the study (three years).
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | GORE VIABAHN Endoprosthesis | Bare Nitinol Stent
Number analyzed (Participants) | 72 | 76
percentage of subjects | 24.2 [12.2 to 38.5] | 25.9 [10.3 to 45.0]

2. Primary Outcome: Safety: Composite of Major Procedural (30-day) Adverse Events (AEs)
Description: Major procedural events include death, myocardial infarction, acute renal insufficiency, study limb amputation, and access site and treatment site complications requiring surgery or blood transfusion. The results for this outcome measure are the total percent of these events that occurred in each treatment arm within the first 30 days following stent implantations.
Time Frame: 30 days
Measure: Number; unit: percentage of subjects
Arm/Group | GORE VIABAHN Endoprosthesis | Bare Nitinol Stent
Number analyzed (Participants) | 72 | 76
percentage of subjects | 1.4 | 0

3. Secondary Outcome: Primary Assisted Patency
Description: Primary assisted patency is defined as when the subject had a repeat intervention to regain patency in order to salvage the stent prior to complete occlusion.
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | GORE VIABAHN Endoprosthesis | Bare Nitinol Stent
Number analyzed (Participants) | 72 | 76
percentage of subjects | 69.8 [53.5 to 81.3] | 88.8 [78.0 to 94.5]

4. Secondary Outcome: Secondary Patency
Description: Secondary patency is defined as maintaining patency in the target vessel after a repeat intervention to correct complete occlusion in the treated arterial segment.
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | GORE VIABAHN Endoprosthesis | Bare Nitinol Stent
Number analyzed (Participants) | 72 | 76
percentage of subjects | 79.5 [62.6 to 89.4] | 89.3 [77.7 to 95.1]

5. Secondary Outcome: Technical Success at Initial Procedure
Description: Technical success is defined as a composite of both a) restoration of superficial femoral artery (SFA) patency with < 30% residual stenosis (narrowing) within the treated arterial segment as viewed on post-procedure completion angiography, and b) Final Hemodynamic Pressure Gradient ≤15mm Hg (mercury). A lower pressure gradient number indicates less resistance to blood flow; i.e., less stenosis or narrowing of the vessel under the pressure of the flow.
  The results show the percentage of study subjects that had technical success.
Time Frame: Time of implant procedure
Population: The number of participant analyzed were those for which we had data. Not all sites recorded both measures required to calculate technical success.
Measure: Number; unit: percentage of subjects
Arm/Group | GORE VIABAHN Endoprosthesis | Bare Nitinol Stent
Number analyzed (Participants) | 69 | 69
percentage of subjects | 97.3 | 85.7

6. Secondary Outcome: Target Vessel Revascularization (TVR)
Description: This measure shows the percentage of subjects that had at least one repeat intervention performed during their enrollment in the clinical study.
Time Frame: 3 years
Measure: Number; unit: percentage of participants
Arm/Group | GORE VIABAHN Endoprosthesis | Bare Nitinol Stent
Number analyzed (Participants) | 72 | 76
percentage of participants | 37.5 | 35.5

7. Secondary Outcome: Target Lesion Revascularization (TLR)
Description: This measure shows the percentage of subjects that had at least one repeat intervention in the target lesion during their enrollment in the clinical study.
Time Frame: 3 years
Measure: Number; unit: percentage of participants
Arm/Group | GORE VIABAHN Endoprosthesis | Bare Nitinol Stent
Number analyzed (Participants) | 72 | 76
percentage of participants | 34.7 | 34.2

8. Secondary Outcome: Improvement in Rutherford Classification (Clinical Success)
Description: The Rutherford Classification is a system used to score Peripheral Artery Disease (PAD). The stages follow (higher numbers are worse):
  Stage 0 - Asymptomatic Stage 1 - Mild claudication Stage 2 - Moderate claudication Stage 3 - Severe claudication Stage 4 - Rest pain Stage 5 - Ischemic ulceration not exceeding ulcer of the digits of the foot Stage 6 - Severe ischemic ulcers or frank gangrene
  The percentage of people improving by at least one stage (moving frm higher number to lower number) is listed in the results.
Time Frame: 3 years
Population: The number of participants analyzed was the number of subjects that returned for the 3yr follow-up visit and for which we had data.
Measure: Number; unit: percentage of participants
Arm/Group | GORE VIABAHN Endoprosthesis | Bare Nitinol Stent
Number analyzed (Participants) | 45 | 48
percentage of participants | 86.7 | 91.7

9. Secondary Outcome: Quality of Life Subject Self-assessments (Intermittent Claudication Questionnaire: ICQ) (Clinical Success)
Description: The ICQ is a series of 16 questions asking about leg pain and limitations to activities such as walking specific distances, doing daily activities, worrying about pain, resting during activities, and similar. Most questions specifically ask about only the two weeks prior to answering the completion of the questionnaire.
  Improvement in Intermittent Claudication Questionnaire (ICQ) is a lower score (0 = best, 100 = worst). A decrease in mean score from baseline indicates an improvement in the patient's condition and an increase indicates a decline.
Time Frame: 3 years
Population: Number of subjects that returned for 3yr follow-up appointment and completed the ICQ.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | GORE VIABAHN Endoprosthesis | Bare Nitinol Stent
Number analyzed (Participants) | 40 | 45
Score
  Baseline | 46.6 (20.1) [8 to 91] | 50.1 (18.2) [8 to 80]
  36month | 20.8 (19.6) | 22.9 (21.2)

10. Secondary Outcome: Quality of Life Subject Self-assessments (Short Form:36 (SF:36) - Mental Summary Score)) (Clinical Success)
Description: The SF-36 Health Survey (version 2) asks 36 questions to measure health and well-being from the patient's point of view. The subscale and total score ranges from 0 to 100 but is normalized so that a score of 50 is the population mean, with a standard deviation of 10.
  The SF:36 - Mental Summary Score Questionnaire score must improve in order to be considered for clinical success. An increase in the mean score from baseline indicates an improvement in the patient's condition and a decrease indicates a decline.
Time Frame: 3 years
Population: The number of participants analyzed is the number of subjects that returned for the 3yr follow-up and completed the assessment.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | GORE VIABAHN Endoprosthesis | Bare Nitinol Stent
Number analyzed (Participants) | 39 | 45
Score
  Baseline mean score | 50.3 (12.8) | 48.3 (11.6)
  36-month Mean | 54 (9.1) | 54 (8.6)

11. Secondary Outcome: Quality of Life Subject Self-assessments (Short Form:36 (SF:36) - Physical Summary Score)) (Clinical Success)
Description: The SF-36 Health Survey (version 2) asks 36 questions to measure health and well-being from the patient's point of view. The subscale and total score ranges from 0 to 100 but is normalized so that a score of 50 is the population mean, with a standard deviation of 10.
  The SF:36 - Physical Summary Score Questionnaire score must improve in order to be considered for clinical success. An increase in the mean score from baseline indicates an improvement in the patient's condition and a decrease indicates a decline.
Time Frame: 3 years
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | GORE VIABAHN Endoprosthesis | Bare Nitinol Stent
Number analyzed (Participants) | 39 | 45
Score
  Baseline Mean | 33.6 (9.9) [14 to 59] | 32.9 (8.5) [14 to 51]
  36-month Mean | 41.9 (11.7) [21 to 61] | 38.7 (10.5) [16 to 59]

12. Secondary Outcome: Change in Ankle-Brachial Index (ABI)
Description: This test is done by measuring blood pressure at the ankle and the arm while a person is at rest. The ABI is then calculated by dividing the systolic blood pressure at the ankle by the systolic blood pressures in the arm.
  A normal resting ABI is 0.9 to 1.3. A resting ABI of less than 0.9 is abnormal.
  An outcome of a higher mean ABI is considered a success.
Time Frame: 3 years
Population: The number of participants analyzed is the number of subjects that returned for the 3yr follow-up and had the ABI completed and recorded.
Measure: Mean (Standard Deviation); unit: ABI Value
Arm/Group | GORE VIABAHN Endoprosthesis | Bare Nitinol Stent
Number analyzed (Participants) | 46 | 44
ABI Value
  Baseline Mean | 0.64 (0.15) | 0.67 (0.16)
  36-month Mean | 0.95 (0.18) | 0.97 (0.16)

13. Secondary Outcome: Alternate Peak Systolic Velocity Ratio (PSVR) (Equal or Less Than 2.5)
Description: The PSVR is the ratio of the highest velocity (or pressure) of the blood moving through the stent divided by the velocity immediately outside the stent (the end of the stent nearest to the heart). Pressures are measured by ultrasound. These results include the percentage of subjects that had a PSVR of equal or less than 2.5.
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | GORE VIABAHN Endoprosthesis | Bare Nitinol Stent
Number analyzed (Participants) | 72 | 76
percentage of subjects | 27.2 [14.1 to 42.0] | 28.6 [13.3 to 46.0]

14. Secondary Outcome: Alternate Peak Systolic Velocity Ratio (Less Than or Equal to 3.0)
Description: The PSVR is the ratio of the highest velocity (or pressure) of the blood moving through the stent divided by the velocity immediately outside the stent (the end of the stent nearest to the heart). Pressures are measured by ultrasound. These results include the percentage of subjects that had a PSVR of equal or less than 3.0.
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | GORE VIABAHN Endoprosthesis | Bare Nitinol Stent
Number analyzed (Participants) | 72 | 76
percentage of subjects | 31.3 [17.4 to 46.2] | 29.2 [11.0 to 50.4]

15. Secondary Outcome: Occurrence of Stent Fracture
Description: The outcome of stent fracture measures the percentages of subjects that had stent fractures, as observed in their 1yr follow-up visit X-rays.
Time Frame: 1 year
Population: The number of participants analyzed is the number of subjects that returned for the 1yr follow-up and completed the X-ray assessment.
Measure: Number; unit: percentage of particpants
Arm/Group | GORE VIABAHN Endoprosthesis | Bare Nitinol Stent
Number analyzed (Participants) | 47 | 55
percentage of particpants | 2.1 | 32.7

16. Secondary Outcome: Occurrence of Stent Fracture
Description: The outcome of stent fracture measures the percentages of subjects that had stent fractures, as observed in their 2yr follow-up visit X-rays.
Time Frame: 2 years
Population: The number of participants analyzed is the number of subjects that returned for the 2yr follow-up and completed the X-ray assessment.
Measure: Number; unit: percentage of participants
Arm/Group | GORE VIABAHN Endoprosthesis | Bare Nitinol Stent
Number analyzed (Participants) | 43 | 47
percentage of participants | 4.7 | 48.9

17. Secondary Outcome: Occurrence of Stent Fracture
Description: The outcome of stent fracture measures the percentages of subjects that had stent fractures, as observed in their 3yr follow-up visit X-rays.
Time Frame: 3 years
Population: The number of participants analyzed is the number of subjects that returned for the 3yr follow-up and completed the X-ray assessment.
Measure: Number; unit: percentage of participants
Arm/Group | GORE VIABAHN Endoprosthesis | Bare Nitinol Stent
Number analyzed (Participants) | 38 | 42
percentage of participants | 2.6 | 50.0

ADVERSE EVENTS:
Time Frame: Throughout three-year study
Description: At each scheduled and unscheduled visit, subjects were asked about their health and if there were any changes to baseline. If so, this was recorded on a Case Report Form and reported to the Sponsor.
Groups:
- GORE VIABAHN Endoprosthesis: GORE VIABAHN Endoprosthesis
- Bare Nitinol Stent: Bare Nitinol Stent
Arm/Group | GORE VIABAHN Endoprosthesis | Bare Nitinol Stent
Serious Adverse Events (participants affected / at risk) | 25/72 | 24/76
Other Adverse Events (participants affected / at risk) | 6/72 | 4/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GORE VIABAHN Endoprosthesis (N=72) | Bare Nitinol Stent (N=76)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Acute chest pain (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiomyopathy NOS (Cardiac disorders) | 1 (1) | 0 (0)
Chest burning (Cardiac disorders) | 0 (0) | 1 (1)
Congestive cardiac failure aggravated (Cardiac disorders) | 0 (0) | 1 (2)
Congestive heart failure (Cardiac disorders) | 3 (4) | 1 (2)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Hypertensive heart disease (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (3) | 1 (1)
Non-Q wave MI (Cardiac disorders) | 1 (1) | 0 (0)
Pulmonary edema (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
GI bleed (Gastrointestinal disorders) | 1 (1) | 0 (0)
Internal hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute chest pain (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Device malfunction (General disorders) | 1 (1) | 0 (0)
Implantable defibrillator malfunction (General disorders) | 0 (0) | 1 (1)
Thrombosis in device (General disorders) | 1 (1) | 0 (0)
Acute bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Acute gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Acute pyelonephritis (Infections and infestations) | 0 (0) | 1 (2)
Bronchitis NOS (Infections and infestations) | 1 (1) | 0 (0)
Candida oesophagitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis gangrenous (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis of foot (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis of hand (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis of leg (Infections and infestations) | 0 (0) | 1 (1)
Influenza A virus infection (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis NOS (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 (0) | 1 (1)
Septicemia due to Escherichia coli (E. coli) (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal septicemia (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision site infection (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Back pain (with radiation) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Calf pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Low back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar vertebral fracture L2 (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain of lower extremities (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bladder cancer NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small cell carcinoma of the lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 1 (1)
Subarachnoid hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Unilateral carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Acute renal insufficiency (Renal and urinary disorders) | 0 (0) | 1 (2)
Chronic renal insufficiency (Renal and urinary disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
AV fistula creation (Surgical and medical procedures) | 0 (0) | 1 (1)
Enucleation of eyeball (Surgical and medical procedures) | 1 (1) | 0 (0)
Claudication (Vascular disorders) | 2 (2) | 3 (3)
Coronary artery disease (Vascular disorders) | 1 (1) | 0 (0)
Coronary heart disease (Vascular disorders) | 1 (1) | 0 (0)
Critical limb ischemia (Vascular disorders) | 1 (1) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
In-stent arterial restenosis (Vascular disorders) | 1 (1) | 0 (0)
Intermittent claudication (Vascular disorders) | 1 (1) | 0 (0)
Ischemic ulcer (Vascular disorders) | 1 (1) | 0 (0)
Leg ischemia (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Superficial femoral arterial stenosis (Vascular disorders) | 1 (1) | 0 (0)
Vessel puncture site thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GORE VIABAHN Endoprosthesis (N=72) | Bare Nitinol Stent (N=76)
Vessel puncture site hematoma (General disorders) | 3 (3) | 1 (1)
Claudication (Vascular disorders) | 4 (8) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator will provide the materials to the sponsor at least 30 days in advance of submission for publication or public disclosure. The sponsor has the right to make modifications as necessary to protect proprietary information or correct inaccuracies in technical specifications or device descriptions.